CLINICAL TRIAL: NCT00818948
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AMG 811 in Subjects With Systemic Lupus Erythematosus With and Without Glomerulonephritis
Brief Title: Safety Study of AMG 811 in Subjects With Systemic Lupus Erythematosus With and Without Glomerulonephritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20070283
Record Dates: First submitted 2008-12-18; First posted 2009-01-08 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-08

CONDITIONS: Nephritis; Systemic Lupus Erythematosus
Keywords: Lupus; Nephritis
MeSH Terms: conditions — Nephritis; Lupus Erythematosus, Systemic | interventions — AMG 811

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 2 subjects of each cohort (cohort 1 to 6) will receive placebo
  Interventions: Drug: AMG 811
- AMG811 (Other): Six subjects in each cohort (cohort 1 to 6) will receive AMG 811
  Interventions: Drug: AMG 811

INTERVENTIONS:
Drug: AMG 811 — Part A of the study will enroll SLE without GN (non-renal) subjects into 3 cohorts (6 AMG 811: 2 placebo). All subjects will receive a dose of AMG 811 or placebo every 4 weeks beginning with day 1 (D1) for a total of 3 injections. Subjects will be followed through to study day 197, 5 months from the last dose of study medication. Part B of the study will enroll SLE subjects with GN into Cohorts 4, 5 and 6 (6 AMG 811: 2 placebo). Similar to Part A, subjects in Cohorts 4, 5 and 6 will be dosed every 4 weeks with AMG 811 or placebo for a total of 3 injections followed by a 5 month follow-up period. For Cohort 6, subjects will be followed by a 6 month follow-up period.

SUMMARY:
This is a 2-part, multi-center, randomized, double-blind, placebo-controlled, multiple dose escalation study, enrolling approximately 48 subjects. Part A of the study will enroll subjects with Systemic Lupus Erythematosus (SLE) without Glomerulonephritis (GN) into 3 cohorts. Part B of the study will enroll SLE subjects with GN into 3 cohorts. The purpose of the study is to evaluate the multiple dose of AMG 811 on safety. Tolerability and pharmacokinetics.

DETAILED DESCRIPTION:
Part A of the study will enroll SLE without GN (non-renal) subjects into 3 cohorts (6 AMG 811: 2 placebo). All subjects will receive a dose of AMG 811 or placebo every 4 weeks beginning with Day 1 (D1) for a total of 3 injections. Subjects will be followed through to study day 197, 5 months from the last dose of study medication.

Part B of the study will enroll SLE subjects with GN into Cohorts 4, 5, and 6 (6 AMG 811: 2 placebo). Similar to Part A, subjects in Cohorts 4, 5, and 6 will be dosed every 4 weeks with AMG 811 or placebo for a total of 3 injections followed by a 5 month follow-up period. For Cohort 6, subjects will be followed by a 6 month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, between the ages of 18 and 70 years of age;
* Body mass index from 18 to 40 kg/m2 [Body Weight (kg)/Height2 (m2)] at screening;
* Diagnosis of SLE at least 6 months before randomization, including a positive antinuclear antibodies (ANA) during screening; if screening ANA is negative, documented historical ANA with a titer of at least 1:80 will be acceptable;
* Any concurrent SLE pharmacologic regimen (including mycophenolate mofetil, azathioprine, leflunomide, methotrexate, and anti-malarials) must be stable for at least 30 days before randomization;
* Prednisone ≤ 20 mg/day (or equivalent) is permitted; one increase or one decrease of ≤ 5 mg/day prednisone equivalent will be allowed within 30 days before randomization;

Additional inclusion criteria for Part B:

- Active SLE with GN with no other apparent cause, defined by the following: Renal biopsy evidence (within 18 months) of nephritis using the WHO or International Society of Nephrology (ISN)/Renal Pathology Society (RPS) classification of SLE with GN (Class III or IV); Urine protein/creatinine ratio (UP/Cr) > 1 or 24 hour urine protein > 1g after at least 12 weeks of treatment with mycophenolate mofetil (at least 1.5 grams/day) or azathioprine (at least 100 mg orally per day); Superimposed membranous changes are allowed for those with Class III or Class IV SLE with GN;

- Prednisone ≤ 20 mg/day (or equivalent) at the time of randomization.

Exclusion Criteria:

* Any disorder (including psychiatric), condition or clinically significant disease (other than a diagnosis of SLE) that would, by its progressive nature and/or severity, interfere with the study evaluation, completion and/or procedures per the investigator's discretion;
* Creatinine clearance within the screening period of less than 50 mL/min as calculated by the Cockcroft-Gault method
* Signs or symptoms of a viral, bacterial or fungal infection within 30 days of study randomization, or recent history of repeated infections;
* Underlying condition other than SLE or being on allowed immunosuppressants that predisposes one to infections
* Prior use of the following agents:
* Administration of an investigational biologic agent that primarily targets the immune system
* Administration of cyclosporine, tacrolimus, sirolimus, IV immunoglobulin, and/or plasmapheresis within 3 months of randomization;
* Administration of oral or IV cyclophosphamide (or any other alkylating agent) within 12 months (Part A) or 3 months (Part B) of randomization;
* History of ethanol or drug abuse within the last one year prior to randomization;

Additional exclusion criteria for Part B:

* Rapidly progressive GN (defined as a doubling of serum creatinine within the past 3 months);
* Evidence of significant chronicity, defined as:

> 50% glomeruli with sclerosis or > 50% interstitial fibrosis on renal biopsy; or International Society of Nephrology (ISN)/Renal Pathology Society (RPS) 2003 Class III (C), IV-S (C) or IV-G (C).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-03; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Safety evaluation: Subject incidence of treatment-emergent adverse events, clinically significant changes in vital signs, physical examination endpoints, clinical laboratory safety tests, ECGs and the development of anti-AMG811 antibodies | 197 days

SECONDARY OUTCOMES:
Serum and urine PK parameters of AMG 811 | 197 days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (12):
- United States (8):
  - Research Site, Phoenix, Arizona
  - Research Site, Danbury, Connecticut
  - Research Site, Kansas City, Kansas
  - Research Site, Manhasset, New York
  - Research Site, New York, New York
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Amarillo, Texas
  - Research Site, Dallas, Texas
- Research Site, Paris, France
- Research Site, Hong Kong, Hong Kong
- Research Site, Kuala Lumpur, Kuala Lumpur, Malaysia
- Research Site, Mexico City, Mexico City, Mexico

REFERENCES:
- [Derived] Boedigheimer MJ, Martin DA, Amoura Z, Sanchez-Guerrero J, Romero-Diaz J, Kivitz A, Aranow C, Chan TM, Chong YB, Chiu K, Wang C, Sohn W, Arnold GE, Damore MA, Welcher AA, Sullivan BA, Kotzin BL, Chung JB. Safety, pharmacokinetics and pharmacodynamics of AMG 811, an anti-interferon-gamma monoclonal antibody, in SLE subjects without or with lupus nephritis. Lupus Sci Med. 2017 Sep 14;4(1):e000226. doi: 10.1136/lupus-2017-000226. eCollection 2017. PMID 29018537
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com